CLINICAL TRIAL: NCT05897307
Title: Dexmedetomidine Ropivacaine Versus Plain Ropivacaine in Bilateral Pectoralis Nerve Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fayoum University Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Hamed, the head of anesthesia department, Fayoum University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: E-23
Record Dates: First submitted 2023-05-23; First posted 2023-06-09 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Post Operative Pain
Keywords: cardiac surgery; fast track anesthesia; postoperative analgesia
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group (C) (Placebo Comparator): will not receive any regional anesthesia and only will receive fentanyl 1μg/kg/hr.
  Interventions: Drug: Ropivacaine
- Group (R) (Active Comparator): will receive 30 ml of 0.25% of plain ropivacaine for each side.
  Interventions: Drug: Ropivacaine
- Group (DR) (Active Comparator): will receive 30 ml of 0.25% of ropivacaine + dexmedetomidine 0.5 μg/kg for each side.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — dexmedetomidine

SUMMARY:
Background: Multimodal analgesia for control of postoperative pain in cardiac surgical patients helps in early recovery and ambulation. Pectoral nerve (PECS) block with ropivacaine is novel, less invasive regional analgesic technique with an effect comparable to paravertebral, and thoracic epidural analgesia.

Aim: The aim of this study is to assess the effect of dexmedetomidine as an adjuvant to ropivacaine on the quality and efficiency of the ultra-sound guided pectoralis nerve block in patients undergoing open heart surgery through midline sternotomy for fast-track anesthesia and postoperative analgesia.

DETAILED DESCRIPTION:
In 2012 Blanco et al. [1] described the ultrasound technique for Pectoral nerve (PECS) block as a new, less invasive regional analgesic technique for breast surgeries.

PECS block includes PECS I and PECS II (modified PECS I) interfascial blocks. Since that time, PECS block has been used successfully with good results for a wide variety of surgeries on chest wall such as radical mastectomies, breast-conserving surgeries, breast implant placement, automated implantable cardioverter-defibrillator (AICD)/pacemaker placement, intercostal drainage tube placement, and rib fractures. [1] PECS I & II blocks are considered very safe due to the lack of major neurovascular bundles surrounding the area of interest [2, 3].

In 2018 Kumar et al. [4] investigated the efficacy of ultrasound-guided bilateral PECS block for patients undergoing cardiac surgery through midline sternotomy approach. They concluded that Pecs block is technically simple, safe, and very effective technique and can be used as a part of multimodal analgesia in postoperative cardiac surgical patients for better patient comfort and satisfaction and also helps in superior pulmonary rehabilitation, thus assisting in better outcome. [4] With ultrasound guidance, this block has a short learning curve, and because it is superficial block, it is easier to apply, and this is one of the reasons for its increasing use and importance, and it is often performed instead of thoracic epidural block (TEA) and thoracic paravertebral block (TPVB). [4] The current data clearly demonstrates earlier extubation and reduced perioperative narcotic consumption [4-6], which are inherently beneficial for the patient. Adequate pain control is critical for respiratory mechanics and metabolic activity, especially for cardiac patients.

Compared with other regional anesthesia techniques, the ability to perform PECS block in the supine position is a critical advantage as it is convenient to place and should not impact the logistics of the operating room workflow. In addition, it has great potential as a postop analgesic option for cardiac surgeries, possibly as a rescue block. [4] Ropivacaine is a long-acting local anaesthetic agent that is less lipophilic than bupivacaine, and this reduced lipophilicity is associated with decreased potential for central nervous system toxicity and cardiotoxicity. [7] Dexmedetomidine is a potent and highly selective α2-adrenoreceptor agonist. It has sedative-hypnotic, anxiolytic, analgesic, anesthetic-reducing and local anesthetic effects. [8] The mechanism of action of dexmedetomidine for potentiation of local anesthetics may be through its central action, α-2 receptor-mediated vasoconstriction, attenuation of inflammatory responses, direct effect on peripheral nerves, or by increasing the activity-dependent hyperpolarization through blocking the hyperpolarization-activated cation (Ih) current. [9] The available preclinical and clinical data propose that the addition of dexmedetomidine with local anesthetics is well tolerated without signs of neurotoxicity. [10] In this study, we hypothesized that adding dexmedetomidine as an adjuvant to ropivacaine can result in prolongation of duration of anesthesia with improvement of the quality of postoperative analgesia of bilateral PECS block for patients undergoing cardiac surgery via midline sternotomy compared with using only plain ropivacaine.

Patients and Methods:

After approval of our local ethical committee, and based upon written informed consent, ninety patients, ASA physical statuses III or IV, undergoing either coronary artery bypass grafting (CABG) or valve surgeries through midline sternotomy will be enrolled in the study.

Inclusion criteria:

* Age 20 - 65 years,
* Ejection fraction (EF) > 35%,
* Elective isolated CABG, or Valve surgery

Exclusion criteria:

* Poor left ventricular function with intra-aortic balloon pump support,
* Recent myocardial infarction (last seven days),
* Combined procedure (i.e., CABG + other heart/vascular procedure),
* Emergency surgery, or Redo cases,
* Hepatic or renal failure, creatinine >1.5,
* Patients with hemodynamic instability, preexisting infection at the site of block, allergy to local anesthetics, psychiatric illness, and patients with prolonged postoperative ventilatory course were excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 - 65 years,
* Ejection fraction (EF) > 35%,
* Elective-isolated CABG, or Valve surgery

Exclusion Criteria:

* Poor left ventricular function with intra-aortic balloon pump support,
* Recent myocardial infarction (last seven days),
* Combined procedure (i.e., CABG + other heart/vascular procedure),
* Emergency surgery, or Redo cases,
* Hepatic or renal failure, creatinine >1.5,
* Patients with hemodynamic instability, preexisting infection at the site of block, allergy to local anesthetics, psychiatric illness, and patients with prolonged postoperative ventilatory course were excluded from the study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-08-10 (Estimated); Study Completion 2024-08-20 (Estimated)

PRIMARY OUTCOMES:
the total postoperative opioid consumption | the first 48 hours postoperative
  the total postoperative opioid consumption

SECONDARY OUTCOMES:
Duration of mechanical ventilation | the first 48 hours postoperative
  Duration of mechanical ventilation (day)

CONTACTS AND LOCATIONS:
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
no plane

REFERENCES:
- [Background] Blanco R, Fajardo M, Parras Maldonado T. Ultrasound description of Pecs II (modified Pecs I): a novel approach to breast surgery. Rev Esp Anestesiol Reanim. 2012 Nov;59(9):470-5. doi: 10.1016/j.redar.2012.07.003. Epub 2012 Aug 29. PMID 22939099
- [Background] Ueshima H, Otake H. RETRACTED: Ultrasound-guided pectoral nerves (PECS) block: Complications observed in 498 consecutive cases. J Clin Anesth. 2017 Nov;42:46. doi: 10.1016/j.jclinane.2017.08.006. Epub 2017 Aug 9. No abstract available. PMID 28802149